CLINICAL TRIAL: NCT00414583
Title: Stroke in Young Fabry Patients (sifap1): Frequency of Fabry Disease in an Unselected Group of Young Stroke Patients: an International, Multicentre Prevalence Study
Brief Title: Stroke in Young Fabry Patients (sifap1): Frequency of Fabry Disease in Young Stroke Patients
Acronym: sifap1
Status: Completed | Type: Observational
Sponsor: CENTOGENE GmbH Rostock (Industry)
Collaborators: Shire Human Genetic Therapies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: II PV03/2006
Record Dates: First submitted 2006-12-19; First posted 2006-12-21 (Estimated); Last update posted 2021-04-09 (Actual); Status verified 2020-04

CONDITIONS: Cerebrovascular Accident
Keywords: Cerebrovascular Accident; Cerebrovascular Accident, Acute; CVA (Cerebrovascular Accident); Cerebral Stroke; Stroke, Acute; Cerebrovascular Stroke; Fabry Disease; Anderson-Fabry Disease; Fabry's Disease
MeSH Terms: conditions — Stroke; Fabry Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fabry diagnostic will be done centrally: blood samples will be retained for analysis of a-galactosidase in blood to diagnose an a-galactosidase deficit; in females direct analysis of the gene has to be done since due to the Lyonisation effect a-galactosidase activity might be normal in blood although the patient might suffer from Fabry disease.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observation: all adult patients (18 - 55 years of age) with an acute cerebrovascular event of any etiology
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational study, only laboratory analysis and diagnostic interventions done; no drug tested
  Other Names: only 1 observational group

SUMMARY:
More than one million people in Europe suffer from a stroke every day. Normally older people have a stroke, but also a significant number of younger people between 18 and 55 years. Usually, these cannot be explained by the classical risk factors such as diabetes, overweight and high blood pressure. New studies indicate that in about 1 - 2 % of the younger stroke patients the cause could have been an undiagnosed genetic disease, the so called Fabry disease. The purpose of this study is to determine in a large number of young stroke patients, how many strokes were caused by Fabry Disease.

DETAILED DESCRIPTION:
Aim:

To determine the frequency of Fabry disease in an unselected group of young patients (18 - 55 years of age) with acute cerebrovascular event (CVE)

Fabry disease and stroke:

Rolfs and co-workers have shown a high frequency of Fabry disease in a cohort of patients with cryptogenic stroke (4 % [28/721]) aged between 18 and 55 years. This corresponds to about 1.2 % in the general population of young stroke patients. Therefore the authors stated that Fabry disease must be considered in all cases of unexplained stroke in young patients, especially in cases with the combination of infarction in the vertebrobasilar artery system and proteinuria.

Cryptogenic strokes are cerebrovascular lesions of unknown origin. Clinical and laboratory data show that Fabry disease is itself a risk factor for accelerated atherosclerosis and cardiac and renal disease, which can lead to emboli and hypertension. The pilot-phase started April 2007; the official study started January 2008.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 - 55 years of age) with an acute cerebrovascular event of any etiology defined as patients having an acute ischemic stroke or transient ischemic attack less than 3 months before enrollment into the study
* MRI-scan evidence of associated corresponding brain infarction or hemorrhage, regardless of the duration of symptoms. Alternatively also patients with no signs of stroke in the MRI can be included if a stroke-experienced neurologist has done the initial diagnosis as ischemic stroke, transient ischemic attack or hemorrhage.
* Detailed MRI documentation at admission to entry to the study
* Diagnostic procedures for CVE according to the EUSI recommendations
* Written informed consent from patient or legal representative according to local regulations

Exclusion Criteria:

* Patients being younger than 18 years or older than 55 years of age.
* Acute ischemic stroke or transient ischemic attack longer than 3 months before enrolment into the study
* Diagnosis of the CVE within the last 3 months has been done by a non-neurologist if there is no MRI-scan evidence of associated brain infarction or hemorrhage
* No detailed MRI documentation at admission to entry to the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult patients (18 - 55 years of age) with an acute cerebrovascular event of any etiology defined as patients having an acute ischemic stroke or transient ischemic attack less than 3 months before enrollment into the study
Sampling Method: Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of Fabry disease in the unselected group of young stroke patients | baseline

SECONDARY OUTCOMES:
Classification of stroke subtype in patients identified to have Fabry disease acc. to TOAST criteria, modified Rankin scale, Barthel index and MRI criteria. | baseline

CONTACTS AND LOCATIONS:
Locations (45):
- Austria (5):
  - Universitätsklinikum für Neurologie, Graz
  - Department of Neurology, Universitaetsklinik fuer Neurologie Innsbruck, Innsbruck
  - Wagner-Jauregg Linz, Department of Neurology, Linz
  - Christian-Doppler-Klinik, Department für medizin. Studien, Salzburg
  - Krankenhaus der Barmherzigen Brüder, Abteilung für Neurologie, Vienna
- Belgium (2):
  - Middelheim General Hospital, Dept. of Neurology/Memory Clinic, Antwerp
  - UZ Gasthuisburg Hospital, Leuven
- Department of Neurology, University Hospital Sestre Milosrdnice, Zagreb, Croatia
- Helsinki University Central Hospital, Department of Neurology, Helsinki, Finland
- Hopital Neurologique de Lyon, Service d'urgences Neurovasculaires, Lyon, France
- Department of Neurology, S. Khechinashvili University clinic of Tbilisi state medical university, Tbilisi, Georgia
- Germany (26):
  - Department of Neurology, Kreiskrankenhaus Altenburg, Altenburg
  - Department of Neurology, Klinikum Hohe Warte, Bayreuth
  - Dept. of Neurology, Vivantes Netzwerk für Gesundheit GmbH, Klinikum Neukölln, Berlin
  - Charite Campus Benjamin Franklin, Dept. of Neurology, Berlin
  - Klinikum Bremen Mitte gGmbH, Neurologische Klinik, Bremen
  - Department of Neurology, Allgemeines Krankenhaus Celle, Celle
  - Department of Neurology, Klinikum Chemnitz gGmbH, Chemnitz
  - Department of Neurology, Universitaetsklinikum Carl Gustav Carus, Dresden
  - Heinrich-Heine University Duesseldorf, Dept. of Neurology, Düsseldorf
  - Dept. of Neurology, Johann-Wolfgang-Goethe-Universität, Frankfurt
  - University of Giessen-Marburg Dept. of Neurology, Giessen
  - Department of Neurology, Ernst-Moritz-Arndt-University, Greifswald
  - Dept. of Neurology, Martin-Luther-Universität, Universitätsklinik und Poliklinik für Neurologie, Halle
  - Department of Neurology S10, Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - University of Heidelberg, Department of Neurology, Heidelberg
  - Department of Neurology, Universitaetsklinikum Jena, Jena
  - University Schleswig-Holstein, Dept. of Neurology, Kiel
  - Department of Neurology, Universitaetsklinikum Leipzig, Leipzig
  - Department of Neurology, Universitaetsklinikum Giessen und Marburg GmbH, Marburg
  - Dept. of Neurology, Ökumenisches Hainich Klinikum gGmbH, Mühlhausen
  - Ludwig-Maximilians-University of Munich, Dept. of Neurology, München
  - University of Muenster, Dept. of Neurology, Münster
  - Department of Neurology, Klinik und Poliklinik fuer Neurologie, Regensburg
  - University of Rostock, Department of Neurology, Rostock
  - Department of Neurology, University Tuebingen, Tübingen
  - University of Ulm, Department of Neurology, Ulm
- The Adelaide and Meath Hospital, Department of Neurology, Dublin, Ireland
- Dept. of Neurology, Ospoedale Maggiore Policlinico, Milan, Italy
- Neuromedical Ward, Mater Dei Hospital, Msida, Malta
- Institute of Psychiatry and Neurology, Dept. of Neurology, Warsaw, Poland
- Centro Hospitalar de Lisboa Central, Servico de Neurologia, Lisbon, Portugal
- Department of Neurology, Hospital Universitario La Paz, Madrid, Spain
- United Kingdom (2):
  - Stroke Prevention Research Unit, Dept. of Clinical Neurology, University of Glasgow, Southern General Hospital, Glasgow, Scotland
  - Stroke Prevention Research Unit, John Radcliffe Hospital, Oxford

REFERENCES:
- [Background] Rolfs A, Bottcher T, Zschiesche M, Morris P, Winchester B, Bauer P, Walter U, Mix E, Lohr M, Harzer K, Strauss U, Pahnke J, Grossmann A, Benecke R. Prevalence of Fabry disease in patients with cryptogenic stroke: a prospective study. Lancet. 2005 Nov 19;366(9499):1794-6. doi: 10.1016/S0140-6736(05)67635-0. PMID 16298216
- [Background] Rolfs A, Martus P, Heuschmann PU, Grittner U, Holzhausen M, Tatlisumak T, Bottcher T, Fazekas F, Enzinger C, Ropele S, Schmidt R, Riess O, Norrving B; sifap1 Investigators. Protocol and methodology of the Stroke in Young Fabry Patients (sifap1) study: a prospective multicenter European study of 5,024 young stroke patients aged 18-55 years. Cerebrovasc Dis. 2011;31(3):253-62. doi: 10.1159/000322153. Epub 2010 Dec 21. PMID 21178350
- [Derived] Thijs V, Grittner U, Fazekas F, McCabe DJH, Giese AK, Kessler C, Martus P, Norrving B, Ringelstein EB, Schmidt R, Tanislav C, Putaala J, Tatlisumak T, von Sarnowski B, Rolfs A, Enzinger C; Stroke in Fabry (SIFAP1) Investigators. Dolichoectasia and Small Vessel Disease in Young Patients With Transient Ischemic Attack and Stroke. Stroke. 2017 Sep;48(9):2361-2367. doi: 10.1161/STROKEAHA.117.017406. Epub 2017 Jul 28. PMID 28754833
- [Derived] Aigner A, Grittner U, Rolfs A, Norrving B, Siegerink B, Busch MA. Contribution of Established Stroke Risk Factors to the Burden of Stroke in Young Adults. Stroke. 2017 Jul;48(7):1744-1751. doi: 10.1161/STROKEAHA.117.016599. Epub 2017 Jun 15. PMID 28619986
- [Derived] von Sarnowski B, Schminke U, Grittner U, Tanislav C, Bottcher T, Hennerici MG, Tatlisumak T, Putaala J, Kaps M, Fazekas F, Enzinger C, Rolfs A, Kessler C; sifap1 Investigators. Posterior versus Anterior Circulation Stroke in Young Adults: A Comparative Study of Stroke Aetiologies and Risk Factors in Stroke among Young Fabry Patients (sifap1). Cerebrovasc Dis. 2017;43(3-4):152-160. doi: 10.1159/000454840. Epub 2017 Jan 14. PMID 28088807
- [Derived] Huber R, Grittner U, Weidemann F, Thijs V, Tanislav C, Enzinger C, Fazekas F, Wolf M, Hennerici MG, McCabe DJ, Putaala J, Tatlisumak T, Kessler C, von Sarnowski B, Martus P, Kolodny E, Norrving B, Rolfs A; Stroke in Young Fabry Patients (SIFAP) Investigators. Patent Foramen Ovale and Cryptogenic Strokes in the Stroke in Young Fabry Patients Study. Stroke. 2017 Jan;48(1):30-35. doi: 10.1161/STROKEAHA.116.013620. Epub 2016 Nov 29. PMID 27899752
- [Derived] Tatlisumak T, Putaala J, Innila M, Enzinger C, Metso TM, Curtze S, von Sarnowski B, Amaral-Silva A, Jungehulsing GJ, Tanislav C, Thijs V, Rolfs A, Norrving B, Fazekas F, Suomalainen A, Kolodny EH. Frequency of MELAS main mutation in a phenotype-targeted young ischemic stroke patient population. J Neurol. 2016 Feb;263(2):257-262. doi: 10.1007/s00415-015-7969-z. Epub 2015 Nov 14. PMID 26566914
- [Derived] Wolf ME, Grittner U, Bottcher T, Norrving B, Rolfs A, Hennerici MG; sifap1 TM investigators. Phenotypic ASCO Characterisation of Young Patients with Ischemic Stroke in the Prospective Multicentre Observational sifap1 Study. Cerebrovasc Dis. 2015;40(3-4):129-35. doi: 10.1159/000434760. Epub 2015 Jul 25. PMID 26227782
- [Derived] Thijs V, Grittner U, Dichgans M, Enzinger C, Fazekas F, Giese AK, Kessler C, Kolodny E, Kropp P, Martus P, Norrving B, Ringelstein EB, Rothwell PM, Schmidt R, Tanislav C, Tatlisumak T, von Sarnowski B, Rolfs A; Stroke in Fabry Investigators. Family History in Young Patients With Stroke. Stroke. 2015 Jul;46(7):1975-8. doi: 10.1161/STROKEAHA.115.009341. Epub 2015 Jun 2. PMID 26038521
- [Derived] Fazekas F, Enzinger C, Schmidt R, Grittner U, Giese AK, Hennerici MG, Huber R, Jungehulsing GJ, Kaps M, Kessler C, Martus P, Putaala J, Ropele S, Tanislav C, Tatlisumak T, Thijs V, von Sarnowski B, Norrving B, Rolfs A; SIFAP 1 Investigators. Brain magnetic resonance imaging findings fail to suspect Fabry disease in young patients with an acute cerebrovascular event. Stroke. 2015 Jun;46(6):1548-53. doi: 10.1161/STROKEAHA.114.008548. Epub 2015 Apr 21. PMID 25899239
- [Derived] Tanislav C, Kropp P, Grittner U, Holzhausen M, Fazekas F, Jungehulsing GJ, Tatlisumak T, von Sarnowski B, Putaala J, Huber R, Thijs V, Schmidt R, Kaps M, Enzinger C, Dichgans M, Norrving B, Rolfs A. Clinically relevant depressive symptoms in young stroke patients - results of the sifap1 study. Neuroepidemiology. 2015;44(1):30-8. doi: 10.1159/000371389. Epub 2015 Jan 31. PMID 25659436
- [Derived] Kaps M, Grittner U, Jungehulsing G, Tatlisumak T, Kessler C, Schmidt R, Jukka P, Norrving B, Rolfs A, Tanislav C; sifap1 Investigators. Clinical signs in young patients with stroke related to FAST: results of the sifap1 study. BMJ Open. 2014 Nov 7;4(11):e005276. doi: 10.1136/bmjopen-2014-005276. PMID 25380809
- [Derived] Tanislav C, Grittner U, Misselwitz B, Jungehuelsing GJ, Enzinger C, von Sarnowski B, Putaala J, Kaps M, Kropp P, Rolfs A, Tatlisumak T, Fazekas F, Kolodny E, Norrving B. Lessons from everyday stroke care for clinical research and vice versa: comparison of a comprehensive and a research population of young stroke patients. BMC Neurol. 2014 Mar 7;14:45. doi: 10.1186/1471-2377-14-45. PMID 24607068
- [Derived] Fazekas F, Enzinger C, Schmidt R, Dichgans M, Gaertner B, Jungehulsing GJ, Hennerici MG, Heuschmann P, Holzhausen M, Kaps M, Kessler C, Martus P, Putaala J, Ropele S, Tanislav C, Tatlisumak T, Norrving B, Rolfs A; sifap1 Investigators. MRI in acute cerebral ischemia of the young: the Stroke in Young Fabry Patients (sifap1) Study. Neurology. 2013 Nov 26;81(22):1914-21. doi: 10.1212/01.wnl.0000436611.28210.ec. Epub 2013 Nov 1. PMID 24186912
- [Derived] Kropp P, Holzhausen M, Kolodny E, Becker U, Dichgans M, Diez-Tejedor E, Enzinger C, Fazekas F, Fuentes B, Karpinska A, Meyer W, Tanislav C, Bottcher T, Rolfs A; Stroke in Young Fabry Patients (sifap) Investigators. Headache as a symptom at stroke onset in 4,431 young ischaemic stroke patients. Results from the "Stroke in Young Fabry Patients (SIFAP1) study". J Neural Transm (Vienna). 2013 Oct;120(10):1433-40. doi: 10.1007/s00702-013-1014-0. Epub 2013 Jun 9. PMID 23748977
- [Derived] von Sarnowski B, Schminke U, Tatlisumak T, Putaala J, Grittner U, Kaps M, Tobin WO, Kinsella JA, McCabe DJ, Hennerici MG, Fazekas F, Norrving B, Kessler C, Rolfs A; sifap1 investigators. Prevalence of stenoses and occlusions of brain-supplying arteries in young stroke patients. Neurology. 2013 Apr 2;80(14):1287-94. doi: 10.1212/WNL.0b013e31828ab2ed. Epub 2013 Mar 6. PMID 23468548
- [Derived] Rolfs A, Fazekas F, Grittner U, Dichgans M, Martus P, Holzhausen M, Bottcher T, Heuschmann PU, Tatlisumak T, Tanislav C, Jungehulsing GJ, Giese AK, Putaala J, Huber R, Bodechtel U, Lichy C, Enzinger C, Schmidt R, Hennerici MG, Kaps M, Kessler C, Lackner K, Paschke E, Meyer W, Mascher H, Riess O, Kolodny E, Norrving B; Stroke in Young Fabry Patients (sifap) Investigators. Acute cerebrovascular disease in the young: the Stroke in Young Fabry Patients study. Stroke. 2013 Feb;44(2):340-9. doi: 10.1161/STROKEAHA.112.663708. Epub 2013 Jan 10. PMID 23306324
- [Derived] von Sarnowski B, Putaala J, Grittner U, Gaertner B, Schminke U, Curtze S, Huber R, Tanislav C, Lichy C, Demarin V, Basic-Kes V, Ringelstein EB, Neumann-Haefelin T, Enzinger C, Fazekas F, Rothwell PM, Dichgans M, Jungehulsing GJ, Heuschmann PU, Kaps M, Norrving B, Rolfs A, Kessler C, Tatlisumak T; sifap1 Investigators. Lifestyle risk factors for ischemic stroke and transient ischemic attack in young adults in the Stroke in Young Fabry Patients study. Stroke. 2013 Jan;44(1):119-25. doi: 10.1161/STROKEAHA.112.665190. Epub 2012 Nov 13. PMID 23150649
- [Derived] Steinicke R, Gaertner B, Grittner U, Schmidt W, Dichgans M, Heuschmann PU, Tanislav C, Putaala J, Kaps M, Endres M, Schmidt R, Fazekas F, Norrving B, Rolfs A, Martus P, Tatlisumak T, Enzinger C, Jungehulsing GJ. Kidney function and white matter disease in young stroke patients: analysis of the stroke in young fabry patients study population. Stroke. 2012 Sep;43(9):2382-8. doi: 10.1161/STROKEAHA.111.645713. Epub 2012 Jun 21. PMID 22723456
- [Derived] Fellgiebel A, Keller I, Martus P, Ropele S, Yakushev I, Bottcher T, Fazekas F, Rolfs A. Basilar artery diameter is a potential screening tool for Fabry disease in young stroke patients. Cerebrovasc Dis. 2011;31(3):294-9. doi: 10.1159/000322558. Epub 2010 Dec 22. PMID 21196729